CLINICAL TRIAL: NCT02303470
Title: Vigorous Exercise Versus Moderate Exercise to Improve Glucose Metabolism and Metabolic Parameters in Women With Polycystic Ovary Syndrome and Insulin Resistance: A Prospective Randomized Pilot Study
Brief Title: PCOS & Insulin Resistance Exercise Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-14816
Record Dates: First submitted 2014-11-25; First posted 2014-12-01 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance
Keywords: Exercise
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vigorous Exercise (Experimental): High-intensity interval training for 15 minutes daily, 5 days per week for 8 weeks
  Interventions: Behavioral: Vigorous Exercise
- Moderate Exercise (Experimental): Brisk walking for 30 minutes daily, 5 days per week for 8 weeks
  Interventions: Behavioral: Moderate Exercise

INTERVENTIONS:
Behavioral: Vigorous Exercise — High-intensity interval training alternates 30 seconds of vigorous exercise with 30 seconds of low-intensity recovery for a total of 15 minutes.
  Other Names: High-intensity interval training
  Arms: Vigorous Exercise
Behavioral: Moderate Exercise
  Arms: Moderate Exercise

SUMMARY:
This study evaluates the feasibility and metabolic effects of implementing a structured exercise program in women with polycystic ovary syndrome and insulin resistance. Participants will be randomized to either 75 minutes of vigorous exercise or 150 minutes of moderate exercise per week.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder with an incidence of 5-8% in reproductive aged women. PCOS is characterized by a collection of signs and symptoms, and as defined by the 2003 Rotterdam criteria must include two out of the following three characteristics: oligo-ovulation or anovulation, polycystic-appearing ovaries, and clinical or biochemical evidence of elevated androgens.

Women with PCOS are also known to have an increased risk of metabolic disorders, including insulin resistance, obesity, cardiovascular disease, and hyperlipidemia. It is has been shown that many of the sequelae of PCOS can be improved by interventions that reduce insulin levels. Previous research has demonstrated that weight reduction and metformin are beneficial in restoring normal ovulation patterns and fertility and can improve hyperandrogenemia and hyperlipidemia. Studies of the effect of lifestyle modifications in women with PCOS have shown that exercise, alone or in combination with changes in diet, can improve ovulation rates and metabolic parameters, and is associated with reduced incidence of insulin resistance. As such, the care of PCOS patients often includes counseling regarding reducing dietary intake and improvement in physical fitness. However, the type of exercise evaluated was inconsistent between many of these studies and varied in intensity, frequency and duration. Therefore, the exercise needed to achieve health benefits in PCOS is not well defined. The Department of Health and Human Services (DHHS) recommends that all Americans get at least 150 minutes per week of moderate aerobic exercise or at least 75 minutes per week of vigorous aerobic activity to maintain health and fitness for all Americans. A critical unanswered question is whether one of these options (moderate versus vigorous) provides superior benefits to women with PCOS.

High-intensity interval training (HIIT) is a form of exercise that combines short intervals of vigorous exercise with lower intensity recovery periods. HIIT has been used as a training modality for high-performance athletes for over a decade. More recently, it has been studied for therapeutic purposes in adults with cardiovascular disease, obesity, and metabolic syndrome. These data suggest that when compared to moderate exercise, HIIT shows greater improvement in aerobic capacity, maximal oxygen consumption, indices of insulin resistance, hyperglycemia, and lipid profiles. HIIT has also been compared with moderate-intensity exercise in patients with type 2 diabetes and has shown a reduction in hyperglycemia, though the data have been controversial. HIIT has not been studied specifically in patients with PCOS.

Studies employing structured exercise programs often have a high drop-out rate and poor post-study continuation rate. An exercise program that requires a fitness facility or other equipment may create a barrier to patient compliance. Additionally, time constraints are often cited as a reason for patient drop-out. Our goal is to create an effective exercise program that can be completed in or around the home, requiring only 15-30 minutes per day.

Participants will be randomized to either 15 minutes of vigorous exercise (HIIT) or 30 minutes of moderate exercise (brisk walking) to be performed 5 days per week for 8 weeks. Exercise training will be performed by an exercise physiologist and participants will then complete their exercise programs independently, using heart rate monitoring and exercise diaries to record exercise intensity. This study will evaluate the feasibility of these exercise plans in terms of patient compliance and safety. We will also evaluate the effect of short-duration, vigorous exercise versus longer-duration, moderate exercise on secondary outcomes such as insulin resistance and metabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS as defined by the 2003 Rotterdam criteria
* Presence of insulin resistance as defined by HOMA IR (Insulin Resistance) > 2.0 or fasting insulin ≥ 12 milliunits per liter (mU/L)
* Physician judges that patient is in adequate physical condition to complete exercise program

Exclusion Criteria:

* Age <18 years old or >50 years old
* BMI >40 kg/m2
* Current tobacco user
* Presence of the following pre-existing co-morbid conditions: diabetes mellitus type 2, uncontrolled hypertension (>140/90mmHg), cardiovascular disease
* Presence of musculoskeletal injury or disease that would interfere with patient's ability to complete exercise program
* Current pregnancy or planning to attempt to conceive in the next 3 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Drop-out Rate | 8 weeks
  Drop-out rate in each arm as a measure of feasibility
Completed Days of Exercise | 8 weeks
  Percentage of completed days of exercise program in each arm as a measure of feasibility

SECONDARY OUTCOMES:
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Baseline, 4 weeks, 8 weeks
  Change in HOMA-IR (calculated from fasting glucose and insulin levels)
Fasting Insulin | Baseline, 4 weeks, 8 weeks
  Change in fasting insulin level
Total Cholesterol | Baseline, 8 weeks
  Change in total cholesterol level
LDL Cholesterol | Baseline, 8 weeks
  Change in LDL cholesterol level
HDL Cholesterol | Baseline, 8 weeks
  Change in HDL cholesterol level
Triglycerides | Baseline, 8 weeks
  Change in triglyceride level
Psychological Effects (Change in performance on Beck Depression Inventory - Fast Screen) | Baseline, 8 weeks
  Change in performance on Beck Depression Inventory - Fast Screen
Androgens (Change in free/total testosterone) | Baseline, 8 weeks
  Change in free/total testosterone

CONTACTS AND LOCATIONS:
Overall Officials: Heather Huddleston, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Center for Reproductive Health, San Francisco, California, United States

REFERENCES:
- [Background] Teede HJ, Hutchison SK, Zoungas S. The management of insulin resistance in polycystic ovary syndrome. Trends Endocrinol Metab. 2007 Sep;18(7):273-9. doi: 10.1016/j.tem.2007.08.001. Epub 2007 Aug 16. PMID 17698366
- [Background] Hoeger K, Davidson K, Kochman L, Cherry T, Kopin L, Guzick DS. The impact of metformin, oral contraceptives, and lifestyle modification on polycystic ovary syndrome in obese adolescent women in two randomized, placebo-controlled clinical trials. J Clin Endocrinol Metab. 2008 Nov;93(11):4299-306. doi: 10.1210/jc.2008-0461. Epub 2008 Aug 26. PMID 18728175
- [Background] Moran LJ, Pasquali R, Teede HJ, Hoeger KM, Norman RJ. Treatment of obesity in polycystic ovary syndrome: a position statement of the Androgen Excess and Polycystic Ovary Syndrome Society. Fertil Steril. 2009 Dec;92(6):1966-82. doi: 10.1016/j.fertnstert.2008.09.018. Epub 2008 Dec 4. PMID 19062007
- [Background] Palomba S, Giallauria F, Falbo A, Russo T, Oppedisano R, Tolino A, Colao A, Vigorito C, Zullo F, Orio F. Structured exercise training programme versus hypocaloric hyperproteic diet in obese polycystic ovary syndrome patients with anovulatory infertility: a 24-week pilot study. Hum Reprod. 2008 Mar;23(3):642-50. doi: 10.1093/humrep/dem391. Epub 2007 Dec 23. PMID 18158291
- [Background] Vigorito C, Giallauria F, Palomba S, Cascella T, Manguso F, Lucci R, De Lorenzo A, Tafuri D, Lombardi G, Colao A, Orio F. Beneficial effects of a three-month structured exercise training program on cardiopulmonary functional capacity in young women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2007 Apr;92(4):1379-84. doi: 10.1210/jc.2006-2794. Epub 2007 Jan 30. PMID 17264174
- [Background] Laursen PB, Jenkins DG. The scientific basis for high-intensity interval training: optimising training programmes and maximising performance in highly trained endurance athletes. Sports Med. 2002;32(1):53-73. doi: 10.2165/00007256-200232010-00003. PMID 11772161
- [Background] Rognmo O, Hetland E, Helgerud J, Hoff J, Slordahl SA. High intensity aerobic interval exercise is superior to moderate intensity exercise for increasing aerobic capacity in patients with coronary artery disease. Eur J Cardiovasc Prev Rehabil. 2004 Jun;11(3):216-22. doi: 10.1097/01.hjr.0000131677.96762.0c. PMID 15179103
- [Background] Racil G, Ben Ounis O, Hammouda O, Kallel A, Zouhal H, Chamari K, Amri M. Effects of high vs. moderate exercise intensity during interval training on lipids and adiponectin levels in obese young females. Eur J Appl Physiol. 2013 Oct;113(10):2531-40. doi: 10.1007/s00421-013-2689-5. Epub 2013 Jul 4. PMID 23824463
- [Background] Tjonna AE, Lee SJ, Rognmo O, Stolen TO, Bye A, Haram PM, Loennechen JP, Al-Share QY, Skogvoll E, Slordahl SA, Kemi OJ, Najjar SM, Wisloff U. Aerobic interval training versus continuous moderate exercise as a treatment for the metabolic syndrome: a pilot study. Circulation. 2008 Jul 22;118(4):346-54. doi: 10.1161/CIRCULATIONAHA.108.772822. Epub 2008 Jul 7. PMID 18606913
- [Background] Balducci S, Zanuso S, Cardelli P, Salvi L, Bazuro A, Pugliese L, Maccora C, Iacobini C, Conti FG, Nicolucci A, Pugliese G; Italian Diabetes Exercise Study (IDES) Investigators. Effect of high- versus low-intensity supervised aerobic and resistance training on modifiable cardiovascular risk factors in type 2 diabetes; the Italian Diabetes and Exercise Study (IDES). PLoS One. 2012;7(11):e49297. doi: 10.1371/journal.pone.0049297. Epub 2012 Nov 21. PMID 23185314
- [Background] Shaban N, Kenno KA, Milne KJ. The effects of a 2 week modified high intensity interval training program on the homeostatic model of insulin resistance (HOMA-IR) in adults with type 2 diabetes. J Sports Med Phys Fitness. 2014 Apr;54(2):203-9. PMID 24509992
- [Background] Hoeger KM, Kochman L, Wixom N, Craig K, Miller RK, Guzick DS. A randomized, 48-week, placebo-controlled trial of intensive lifestyle modification and/or metformin therapy in overweight women with polycystic ovary syndrome: a pilot study. Fertil Steril. 2004 Aug;82(2):421-9. doi: 10.1016/j.fertnstert.2004.02.104. PMID 15302293
- [Background] Tanaka H, Monahan KD, Seals DR. Age-predicted maximal heart rate revisited. J Am Coll Cardiol. 2001 Jan;37(1):153-6. doi: 10.1016/s0735-1097(00)01054-8. PMID 11153730
- [Derived] Wang A, Noel M, Christ JP, Corley J, Lenhart N, Cedars MI, Huddleston H. Vigorous vs. moderate exercise to improve glucose metabolism in inactive women with polycystic ovary syndrome and insulin resistance: a pilot randomized controlled trial of two home-based exercise routines. F S Rep. 2023 Dec 22;5(1):80-86. doi: 10.1016/j.xfre.2023.12.004. eCollection 2024 Mar. PMID 38524210